CLINICAL TRIAL: NCT04032314
Title: Lower Extremity Outcome Measures: A Cross-sectional and Longitudinal Observation of Kinematic, Kinetic and Electromyographic Parameters Focussing on Lower Extremity Function in Spinal Cord Injured Patients
Brief Title: Lower Extremity Outcome Measures in SCI
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01451
Record Dates: First submitted 2018-11-13; First posted 2019-07-25 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls - cross-sectional project design
- Patients - cross-sectional project design
- Patients - longitudinal project design

SUMMARY:
Lower extremity (LE) function of patients with a spinal cord injury (SCI) will be assessed in an observational project with a cross-sectional and a longitudinal study design. The main goal is to identify kinematic and kinetic parameters to precisely characterize LE function and in parallel the impairment and limitation in SCI patients throughout rehabilitation in acute patients and in chronic patients to define LE function and LE recovery.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Age 18-80
* Written informed consent
* General consent
* Spinal cord injury (SCI)
* ASIA A-D injury with lowest extent of lesion between C1 and Th12
* Mini-Mental stat examintation score > 26

Exclusion Criteria - Patients:

* Inability to undertake any component of the trial protocol
* Clinically significant conditions such as severe cardiovascular, pulmonary or malignant disease
* Pure cauda equina i.e. peripheral nerve injury

Inclusion Criteria - Healthy controls:

* Age 18-80
* Written informed consent
* General consent

Exclusion Criteria - Healthy controls:

* Reliance on walking aids / prostheses for mobilisation
* Orthopaedic diagnosis with potential impact on gait
* Previous operations on the lower limbs or spine with potential impact on gait
* Inabilitay to undertake any component of the trial protocol
* Clinically significant conditions such as severe cardiovascular, pulmonary or malignant disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an acute or chronic spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Kinematic movement analysis recorded with a motion capture system | Cross-sectional part: one measurement timepoint for patients with chronic SCI within 2 weeks after inclusion (chronic is defined as > 6 months after injury)
  Kinematic movement variables crucial for recovery in lower extremity function after SCI are monitored throughout rehabilitation to generate complex and sensitive profiles of the neurological and functional recovery
Kinematic movement analysis recorded with a motion capture system | Longitudinal part: approx. one measurement timepoint per month where outcome measures will be assessed. Starting < 6 weeks after SCI and continued up to 6 months (or end of rehabilitation).
  Kinematic movement variables crucial for recovery in lower extremity function after SCI are monitored throughout rehabilitation to generate complex and sensitive profiles of the neurological and functional recovery
Kinematic movement analysis recorded with a motion capture system | Longitudinal part: approx. one measurement timepoint per month where outcome measures will be assessed. Starting < 6 weeks after SCI and continued up to 6 months (or end of rehabilitation)
  Kinematic movement variables crucial for recovery in lower extremity function after SCI are monitored throughout rehabilitation to generate complex and sensitive profiles of the neurological and functional recovery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Balgrist, Zurich, Canton of Zurich, Switzerland